CLINICAL TRIAL: NCT07286643
Title: Point-of-care Echocardiogram (POCUS) Guided Resuscitation Versus Conventional Goal- Directed Therapy in the Management of Cirrhosis With Severe Sepsis or Septic Shock: A Randomised Controlled Trial
Brief Title: Echocardiography-guided Cirrhosis and Liver Failure-Intensive Care Protocol Sepsis
Acronym: ECLIPSE-I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGI/IEC/02/2024-3008
Record Dates: First submitted 2024-05-22; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Cirrhosis, Liver; Cirrhotic Cardiomyopathy; Septic Shock
Keywords: echocardiography; cardiac output monitoring; hemodynamics; fluid resuscitation.; POCUS
MeSH Terms: conditions — Liver Cirrhosis; Shock, Septic

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Masking Description: POC ECHO and CGDT Arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECHO arm (Experimental): Other Names: Point of Care- Echo-cardiogram,POCUS Description: • The patients in septic shock with MAP< 65mmHg, with IVC diameter <18mm and IVCCI≥40% in spontaneously breathing patients, would be regarded as fluid depleted state and will be given a fluid challenge with 250-500 ml of balanced salt solution. Those who increment cardiac index by 15% will be continued on fluid boluses with BSS and 5% albumin will be started as ongoing resuscitation within 1 h, which is a standard fluid of choice in patients with cirrhosis soon after the bolus BSS is infused. Fluids will be administered as per periodic POCUS with cardiac US targets, IVC, IJV indices, delta Velocity time integral, and maintenance of MAP>65 mmHg. In the Intervention arm (ECHO) arm, we propose a dynamic Cardiac ultrasound target-based fluid resuscitation strategy.
  Interventions: Diagnostic Test: POCUS
- Conventional goal directed therapy. (CGDT) (Active Comparator): Fixed Target Strategy Fluid boluses would be administered until a central venous pressure (CVP) of 8-10 mmHg is achieved. Till the central line is placed, the shock index (heart rate/ systolic blood pressure) will be used instead of the CVP and IVC indices. Thus fluids (500 ml balanced salt solution followed by 5% albumin) will be administered for a shock index ≥1 and till CVP is placed. • When CVP goal is achieved vasopressors will be started to target MAP ≥ 65mmHg. Once MAP target is achieved, ScVO2 ≥70% and lactate clearance >10% will be targeted. • If ScVO2 is <70% and lactate clearance is <10%, noradrenaline will be started and titrated upwards. take it up to a maximum dose. • Second choice of pressor agent will be vasopressin. • Thus. CGDT group targets CVP, MAP, followed by ScVO2 ≥70% and lactate clearance .
  Interventions: Diagnostic Test: Fixed Resuscitation Strategy based on Target MAP

INTERVENTIONS:
Diagnostic Test: POCUS — * In the Intervention arm (ECHO) arm, we propose a Cardiac ultrasound target-based fluid resuscitation. This incorporates the fluid assessment based on POCUS and myocardial dysfunction based on cardiac ultrasound (cardiac index, myocardial contractility, stroke volume) and portal hypertension-related systemic vasodilation accentuated by sepsis (systemic vascular resistance index or SVRI).
  * The POCUS -velocity time integral and stroke volume index will be used to determine fluid responsiveness.
  * If there is an increment in cardiac index by 15% after giving a fluid bolus (i.e. 250-500 ml of BSS in 15min), we can define 'fluid responsiveness' present.
  * The achievement of lactate clearance, MAP target >65mmHg and ScV02 >70% remains similar as the fixed target strategy.
  The main resuscitation fluid remains 5% albumin in this arm. Albumin infusion will be titrated based on lung ultrasound.
  Arms: ECHO arm
Diagnostic Test: Fixed Resuscitation Strategy based on Target MAP — • Fluid boluses would be administered until a CVP of 8-10 mmHg is achieved and IVC diameter is between 1.8-2 cm with 20-30% collapsibility.
  Till the central line is placed, the shock index (heart rate/ systolic blood pressure) will be used instead of the CVP. Thus fluids (500 ml crystalloid followed by 5% albumin) will be administered for a shock index ≥1 and till CVP is placed.
  * When CVP goal is achieved vasopressors will be started to target MAP ≥ 65mmHg. Once MAP target is achieved, ScVO2 ≥70% and lactate clearance >10% will be targeted.
  * If ScVO2 is <70% and lactate clearance is <10%, noradrenaline will be started and titrated upwards. take it up to a maximum dose.
  * Second choice of pressor agent will be vasopressin.
  * Thus. CGDT group targets CVP, MAP>65 mmHg, followed by ScVO2 ≥70% and lactate clearance in a step wise way.
  Arms: Conventional goal directed therapy. (CGDT)

SUMMARY:
* Point-of-care echocardiography is used to guide septic shock resuscitation in patients with severe sepsis in the intensive care unit (ICU), but without systematic evidence for efficacy in critically patients with Cirrhosis and Severe Sepsis.
* Due to portal hypertension, these patients have a hyperdynamic circulation, increased capillary permeability, splanchnic arteriolar vasodilation, reduced effective circulating blood volume and may have latent cirrhotic cardiomyopathy (CCM).
* Hence assessment of volume status and cardiac reserve using conventional central venous pressure (CVP) or mean arterial pressure (MAP) remains difficult.

Novelty:

* In two recent trials, the role of 5% albumin vs PlasmalyteTM (FRISC study)(1) and 20% albumin vs. PlasmalyteTM (ALPS study) (2) were reported as the primary resuscitation fluid. Neither trial showed a clear long term survival benefit of albumin over balanced salt solution (BSS). In fact, the ALPS trial reported that there was increased risk of pulmonary edema with use of 20% albumin as fluid resuscitation.
* A major limitation of such trial data is that the focus is on choice of fluid rather than looking at hemodynamic goals of resuscitation, resulting in protocolized overzealous fluid administration.
* This may result in albumin-related pulmonary edema, and precipitation of overt heart failure in patients with silent CCM.
* POC-Echo-based fluid resuscitation can prevent pulmonary edema and consequently respiratory failure, while ensuring renal and tissue perfusion.
* It is unclear if choice of fluid or appropriate targets of resuscitation drive the survival benefit in the intensive care management of cirrhosis with severe sepsis.

Objectives:

* The investigators will conduct an ICU based randomised controlled feasibility trial comparing two measures of resuscitation: Echocardiography (ECHO) Guided septic shock resuscitation vs. a modified Goal-Directed Fluid Therapy (GDT) as recommended by sepsis guidelines which use protocol fluids.
* The study will validate the role of POC-Echo parameters as volume assessment tools (cardiac index, systemic vascular resistance index) to determine endpoints of fluid resuscitation and need for vasopressors.
* Lastly, the study aims to determine the presence of CCM in this population, and its impact on clinical outcomes.

Methods POC-ECHO will be done within 1 hours of admission to the liver ICU and at 24h, 48 h and 72 hours in patients with cirrhosis with systolic blood pressure of <90 mmHg or a mean arterial pressure <65 mmHg. Resuscitation target is maintenance of MAP ≥65 mmHg with use of fluids and/or vasopressors. Clinical, cardiac biomarkers, and survival data based on resuscitation fluids will be prospectively collected. CCM will be defined as per CCM Consortium (2020) criteria.

Expected outcome.

The key questions to be answered in the resuscitation of critically ill patients with cirrhosis and sepsis induced hypotension are:

1. What should be best method of ensuring adequate fluid resuscitation i.e. fluid resuscitation protocol?
2. Which measurable clinical parameter can be used to determine adequacy of fluid resuscitation, and as a predictor of mortality outcomes at 7 and 28 days?
3. Whether early fluid resuscitation translates into better clinical outcome in decreasing duration of hospital and intensive care unit (ICU) stay, prevention of AKI and prevention of secondary sepsis?

DETAILED DESCRIPTION:
* Patients with cirrhosis requiring intensive care for severe sepsis carry a risk of high mortality due to altered hemodynamics with reduced effective arterial volume, portal hypertension, presence of ascites, and risk of complications like acute variceal bleeding (AVB), acute kidney injury (AKI) and circulatory failure(3-5). The main principles for management of severe sepsis include early recognition, control of the source of infection, appropriate and timely administration of antimicrobial agents, and resuscitation with intravenous fluids +/- vasoactive drugs, if needed (6).
* Due to portal hypertension, these patients have a hyperdynamic circulation, increased capillary permeability, splanchnic arteriolar vasodilation, and may have latent cirrhotic cardiomyopathy (CCM) (7). Hence assessment of volume status and cardiac reserve using conventional central venous pressure (CVP) or mean arterial pressure (MAP) remains difficult (8). Although inferior vena cava (IVC) dynamics and IVC collapsibility index are reasonable accurate for ventilated patients, their use in spontaneously breathing subjects or those with tense ascites are not defined(9). Even measures like passive leg raising and Valsalva manoeuvre are difficult to perform in cirrhotic patients with tense ascites.
* Early goal directed therapy (EGDT) improved outcomes in a randomized trial in patients with severe sepsis(10). Thereafter EGDT was incorporated into the 6-hour resuscitation bundle of the surviving sepsis campaign guidelines, but did not incorporate patients with cirrhosis(11-13). Following the early EGDT trials, studies focussed choice of resuscitation fluid i.e., albumin versus normal saline or balanced salt solution (BSS), concerns about potential risks of volume overload and pulmonary edema and lack of generalisability in subsequent trials showed that there was no associated survival benefit with an aggressive fluid protocol(14, 15). In the ALBIOS study, 1818 patients with severe sepsis or septic shock were randomized either to receive 300 ml of 20% albumin plus crystalloid or to receive crystalloid alone initially to achieve the EGDT goals. However, no mortality benefit was demonstrated at 29 or 90 days(16).
* Intravenous albumin improves effective circulatory volume by improving plasma oncotic pressure and expands the total blood volume making it the apparent 'fluid of choice' for resuscitation in cirrhosis. The 5% albumin expands plasma volume by 80% of the administered volume, 20% albumin by 210% and 25% albumin by 260% which is expected to remain in the intravascular compartment longer than balanced salt solutions or normal saline(17). In two recent trials, the role of 5% albumin vs PlasmalyteTM (FRISC study) (1)and 20% albumin vs. PlasmalyteTM (ALPS study)(2) were reported as the primary resuscitation fluid. Neither trial showed a clear long term survival benefit of albumin over BSS.
* Point-of-care ultrasonography (POCUS), including cardiac ultrasound, is used to assess volume status, and hemodynamic parameters like cardiac output, systemic vascular resistance, cardiac contractility, and pulmonary artery pressure, which aid in the early and accurate diagnosis of heart failure, cirrhotic cardiomyopathy, porto-pulmonary hypertension, hepatopulmonary syndrome, arrhythmia, pulmonary embolism, and ischemic heart disease. This helps determine the ideal amount of fluids, and vasopressors in resuscitation of patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Critically ill patient with cirrhosis of any etiology
2. Sepsis-related Hypotension (MAP <65mmHg or SBP <90mmHg)
3. 18-65 yrs of age -

Exclusion Criteria:

1. Already on vasopressors/inotropes
2. Severe pre-existing cardiopulmonary disease like porto-pulmonary hypertension (PPH), known coronary artery disease, congenital or valvular heart disease, prosthetic cardiac valves, dilated or restrictive cardiomyopathy.
3. Poor chest wall window due to left pleural effusion, left pneumothorax, small intercostal spaces that restrict performance of a POCUS.
4. Active bleeding like variceal bleed
5. Cerebrovascular events
6. Chronic renal disease - End Stage Renal Disease (ESRD)/ patient on renal replacement therapy
7. Admission to ICU following liver transplantation, burns, cardiac surgery
8. Previous transjugular intra hepatic portosystemic shunt (TIPS),
9. Hepatocellular carcinoma
10. Pregnant or lactating women
11. Informed consent refused by patient or attendants
12. Active COVID-19 infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in volume of resuscitation fluid to attain reversal of shock in POCUS vs Conventional goal-directed therapy at 24 h | Time of randomization to 24 hours
  Dose of balanced salt solution (BSS) and 5% albumin in either arm

SECONDARY OUTCOMES:
Assessment of all-cause mortality | From time of randomization up to Day 7
  Deaths due to liver related or non-liver related causes
Attainment of MAP> 65mmHg | from time of randomization up to time point of reversal of shock
  Assessment of reversal of Shock with attainment of MAP target, and patient being off vasopressors
Assessment of all-cause mortality | From date of randomization until Day 28
Total dose of vasopressor usage in either arm. | From date of randomization until 24 hours
Total dose of vasopressor usage in either arm. | From date of randomization until Day 7
Duration of ICU stay. | From date of randomization until discharge from ICU or death
Cardiac related biomarker panel test | At the Time of Randomization
  NT proBNP, Plasma renin activity and galectin-3.
Cardiac biomarker panel test | The time point of 24 hours from randomization
  Level of NT proBNP, Plasma renin activity and galectin-3.
Cardiac related biomarker panel test | At the Time point of 72h from randomization
  NT proBNP, Plasma renin activity and galectin-3.
Sepsis related biomarker panel test | At the Time of randomization
  sepsis biomarkers procalcitonin, endotoxin, IL-1, IL-6,
Sepsis related biomarker panel test | At the time point of 24 hours from randomization
  sepsis biomarkers procalcitonin, endotoxin, IL-1, IL-6,
Sepsis related biomarker panel test | At the Time point of 72 h from randomization
  sepsis biomarkers procalcitonin, endotoxin, IL-1, IL-6,
Development of any episode of AKI | From randomization till 7 days from enrolment

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No